CLINICAL TRIAL: NCT00555620
Title: A Phase 1 Study Of Sunitinib Malate In Combination With Cisplatin/Capecitabine Or Oxaliplatin/Capecitabine In Patients With Advanced Gastric Cancer
Brief Title: Study Of Sunitinib In Combination With Cisplatin/Capecitabine Or Oxaliplatin/Capecitabine In Patients With Advanced Gastric Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A6181126
Record Dates: First submitted 2007-11-06; First posted 2007-11-08 (Estimated); Results first posted 2011-09-05 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms | interventions — Capecitabine; Oxaliplatin; Sunitinib; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: capecitabine; Drug: oxaliplatin; Drug: sunitinib malate
- B (Experimental)
  Interventions: Drug: capecitabine; Drug: cisplatin; Drug: sunitinib malate

INTERVENTIONS:
Drug: capecitabine — Capecitabine is given orally at 1000mg/m^2 twice a day for 14 days followed by 7 days of drug free period.
  Arms: A
Drug: oxaliplatin — Oxaliplatin is given 110mg/m^2 through a vein on day 1 every 21 days. Each 21 day cycle is repeated until progression of disease or unacceptable toxicity is observed.
  Arms: A
Drug: sunitinib malate — sunitinib is given orally 25mg/day for 14 days followed by 7 days of drug free period.
  Other Names: Sutent
  Arms: A
Drug: capecitabine — Capecitabine is given orally at 1000mg/m^2 twice a day for 14 days followed by 7 days of drug free period.
  Arms: B
Drug: cisplatin — Cisplatin is given 80mg/m^2 through a vein on day 1 every 21 days. Each 21 day cycle is repeated until progression of disease or unacceptable toxicity is observed.
  Arms: B
Drug: sunitinib malate — sunitinib is given orally 25mg/day for 14 days followed by 7 days of drug free period.
  Arms: B

SUMMARY:
The purpose of the study is to determine the safe and tolerable doses of sunitinib given together with either cisplatin and capecitabine or oxaliplatin and capecitabine in patients who have advanced gastric cancer who have not received prior chemotherapy for their advanced cancer

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of stomach cancer
* advanced stomach cancer of stage IV
* adequate blood chemistry, blood counts and kidney function
* willing to participate to study requirements and sign an informed consent document

Exclusion Criteria:

* prior chemotherapy for the stomach cancer in its advanced stage
* excessive toxicities related to prior therapies
* pregnant or breastfeeding patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2008-05; Primary Completion 2010-08 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- South Korea (3):
  - Pfizer Investigational Site, Goyang-si, Gyeonggi-do
  - Pfizer Investigational Site, Seongnam-si, Gyeonggi-do
  - Pfizer Investigational Site, Seoul

REFERENCES:
- [Derived] Lee KW, Park SR, Oh DY, Park YI, Khosravan R, Lin X, Lee SY, Roh EJ, Valota O, Lechuga MJ, Bang YJ. Phase I study of sunitinib plus capecitabine/cisplatin or capecitabine/oxaliplatin in advanced gastric cancer. Invest New Drugs. 2013 Dec;31(6):1547-58. doi: 10.1007/s10637-013-0032-y. Epub 2013 Oct 4. PMID 24091982
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181126&StudyName=Study%20Of%20Sunitinib%20%20In%20Combination%20With%20Cisplatin/Capecitabine%20Or%20Oxaliplatin/Capecitabine%20In%20Patients%20With%20Advanced%20Gastric%20Cancer

RESULTS

PARTICIPANT FLOW:
Groups:
- SU 37.5 mg, CIS 60 mg/m^2, CAP 1600 mg/m^2: Sunitinib (SU): 37.5 milligram (mg) oral capsule daily for 2 weeks (14 days) followed by 1 week (7 days) off treatment (Schedule 2/1). Cisplatin (CIS): 60 mg per meter squared (mg/m^2) intravenous (IV) on Day 1 of each 21-day cycle. Capecitabine (CAP): 800 mg/m^2 oral tablets twice-a-day (BID) on Days 1-14 of each 21-day cycle.
- SU 37.5 mg, CIS 60 mg/m^2, CAP 2000 mg/m^2: SU: 37.5 mg oral capsule Schedule 2/1. CIS: 60 mg/m^2 IV on Day 1 of each 21-day cycle. CAP: 1000 mg/m^2 oral tablets BID on Days 1-14 of each 21-day cycle.
- SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2: SU: 25 mg oral capsule Schedule 2/1. CIS: 80 mg/m^2 IV on Day 1 of each 21-day cycle. CAP: 1000 mg/m^2 oral tablets BID on Days 1-14 of each 21-day cycle.
- SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2: SU: 37.5 mg oral capsule Schedule 2/1. Oxaliplatin (OXA): 110 mg/m^2 IV on Day 1 of each 21-day cycle. CAP: 800 mg/m^2 oral tablets BID on Days 1-14 of each 21-day cycle.
- SU 37.5 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2: SU: 37.5 mg oral capsule Schedule 2/1. OXA: 110 mg/m^2 IV on Day 1 of each 21-day cycle. CAP: 1000 mg/m^2 oral tablets BID on Days 1-14 of each 21-day cycle.
- SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2: SU: 25 mg oral capsule Schedule 2/1. OXA: 110 mg/m^2 IV on Day 1 of each 21-day cycle. CAP: 1000 mg/m^2 oral tablets BID on Days 1-14 of each 21-day cycle.
Period: Overall Study
Arm/Group | SU 37.5 mg, CIS 60 mg/m^2, CAP 1600 mg/m^2 | SU 37.5 mg, CIS 60 mg/m^2, CAP 2000 mg/m^2 | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2
Started | 6 | 7 | 15 | 23 | 3 | 22
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 7 | 15 | 23 | 3 | 22
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Study terminated by sponsor | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 5 | 0 | 1
Not completed — Objective progression or relapse | 6 | 5 | 12 | 17 | 3 | 16
Not completed — Participant refused treatment | 0 | 1 | 1 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 1 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SU 37.5 mg, CIS 60 mg/m^2, CAP 1600 mg/m^2 | SU 37.5 mg, CIS 60 mg/m^2, CAP 2000 mg/m^2 | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2 | Total
Number analyzed (Participants) | 6 | 7 | 15 | 23 | 3 | 22 | 76
Age Continuous [Mean (Standard Deviation); unit: years] | 55.2 (5.8) | 50.0 (12.4) | 50.9 (11.3) | 54.3 (10.1) | 63.3 (11.6) | 50.1 (11.5) | 52.4 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 6 | 6 | 1 | 8 | 23
  Male | 6 | 5 | 9 | 17 | 2 | 14 | 53

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First-cycle Dose Limiting Toxicities (DLTs)
Description: Any DLT event in Cycle 1: Grade (GR) 3/4 nausea, vomiting, or diarrhea despite anti-emetics, anti-diarrheals; GR 3 nonhematological toxicity for greater than or equal to (≥)7 days (except alopecia, skin or hair discoloration, hyperamylasemia, or hyperlipasemia without other clinical evidence of pancreatitis and asymptomatic hyperuricemia); GR 4 nonhematological toxicity; GR 4 neutropenia ≥7 days or thrombocytopenia; GR ≥3 febrile neutropenia or neutropenic infection; GR 3 thrombocytopenia ≥7 days; any treatment-related toxicity having >3 consecutive CAP or SU missed doses per cycle; delayed toxicity recovery >14 days.
Time Frame: Baseline up to Day 21
Population: DLT subpopulation analysis set population: all participants who received at least 1 dose of study drug and did not permanently discontinue during the first cycle of treatment for reasons other than a DLT or miss more than 3 consecutive doses of sunitinib or capecitabine for reasons other than for drug related toxicities within the first cycle.
Measure: Number; unit: participants
Arm/Group | SU 37.5 mg, CIS 60 mg/m^2, CAP 1600 mg/m^2 | SU 37.5 mg, CIS 60 mg/m^2, CAP 2000 mg/m^2 | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2
Number analyzed (Participants) | 6 | 6 | 14 | 21 | 3 | 22
participants | 1 | 0 | 3 | 2 | 2 | 0

2. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of SU, SU012662 (Metabolite of SU), and Total Drug (SU + SU012662)
Time Frame: Day 14 of Cycle 1 (predose and 2, 4, 6, 8, 10, and 24 hours postdose)
Population: Pharmacokinetic (PK) analysis set population: all participants who received sunitinib and had sufficient plasma concentration data to facilitate calculation of the PK parameters; number of participants analyzed (N): participants with evaluable data
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2
Number analyzed (Participants) | 2 | 9 | 10
nanograms per milliliter (ng/mL)
  Cmax SU011248 | 40.1 (10.8) | 69.7 (17.6) | 46.5 (10.8)
  Cmax SU012662 | 14.0 (11.3) | 23.7 (9.9) | 16.6 (3.3)
  Cmax total drug (SU011248+SU012662) | 53.9 (22.1) | 93.0 (24.9) | 62.4 (13.4)

3. Secondary Outcome: Cmax of CAP
Time Frame: Day 1 of Cycle 1 (0.25, 0.5, 1, 2, 3, 4, 8, and 10 hours postdose); Day 14 of Cycle 1 (predose and 0.25, 0.5, 1, 2, 3, 4, 8, and 10 hours postdose)
Population: PK analysis set population; number of participants analyzed (N): participants with evaluable data
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2
Number analyzed (Participants) | 2 | 9 | 10
ng/mL
  Cycle 1, Day 1 | 7000 (7354) | 2051 (1109) | 11681 (8034)
  Cycle 1, Day 14 | 20491 (27098) | 1989 (1686) | 16276 (15832)

4. Secondary Outcome: Cmax of 5'-Deoxy-5-fluorocytidine (Metabolite of CAP, 5'DFCR)
Time Frame: as for outcome 3
Population: PK analysis set population; number of participants analyzed (N): participants with evaluable data
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2
Number analyzed (Participants) | 2 | 9 | 10
ng/mL
  Cycle 1, Day 1 | 4800 (863) | 3352 (1255) | 8017 (3692)
  Cycle 1, Day 14 | 5500 (5982) | 2267 (933) | 8036 (3540)

5. Secondary Outcome: Cmax of 5'-Deoxy-5-fluorouridine (Metabolite of CAP, 5'DFUR)
Time Frame: as for outcome 3
Population: PK analysis set population; number of participants analyzed (N): participants with evaluable data
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2
Number analyzed (Participants) | 2 | 9 | 10
ng/mL
  Cycle 1, Day 1 | 4010 (1909) | 2891 (1099) | 7166 (4073)
  Cycle 1, Day 14 | 6259 (7381) | 2074 (765) | 10082 (5421)

6. Secondary Outcome: Cmax of 5-fluorouracil (Metabolite of CAP, 5-FU)
Time Frame: as for outcome 3
Population: PK analysis set population; number of participants analyzed (N): participants with evaluable data
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2
Number analyzed (Participants) | 2 | 9 | 10
ng/mL
  Cycle 1, Day 1 | 176 (127) | 165 (63) | 495 (326)
  Cycle 1, Day 14 | 552 (641) | 153 (78) | 866 (473)

7. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin) of SU, SU012662, and Total Drug (SU + SU012662)
Time Frame: Day 14 of Cycle 1 (predose and 2, 4, 6, 8, 10, and 24 hours postdose)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2
Number analyzed (Participants) | 2 | 9 | 10
ng/mL
  Cmin SU011248 | 29.0 (5.2) | 49.2 (13.0) | 30.2 (9.2)
  Cmin SU012662 | 11.9 (9.3) | 18.7 (7.9) | 11.1 (2.6)
  Cmin total drug (SU011248+SU012662) | 41.6 (15.6) | 68.5 (16.4) | 41.8 (11.3)

8. Secondary Outcome: Cmin of CAP
Time Frame: as for outcome 3
Population: PK analysis set population; number of participants analyzed (N): participants with evaluable data
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2
Number analyzed (Participants) | 2 | 9 | 10
ng/mL
  Cycle 1, Day 1 | 24.8 (35.1) | 0.0 (0.0) | 0.0 (0.0)
  Cycle 1, Day 14 | 32.0 (45.2) | 0.0 (0.0) | 0.0 (0.0)

9. Secondary Outcome: Cmin of 5'DFCR
Time Frame: as for outcome 3
Population: PK analysis set population; number of participants analyzed (N): participants with evaluable data
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2
Number analyzed (Participants) | 2 | 9 | 10
ng/mL
  Cycle 1, Day 1 | 11.1 (15.7) | 13.0 (20.7) | 55.60 (100.9)
  Cycle 1, Day 14 | 50.5 (71.4) | 0.00 (0.00) | 0.00 (0.00)

10. Secondary Outcome: Cmin of 5'DFUR
Time Frame: as for outcome 3
Population: PK analysis set population; number of participants analyzed (N): participants with evaluable data
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2
Number analyzed (Participants) | 2 | 9 | 10
ng/mL
  Cycle 1, Day 1 | 0.0 (0.0) | 2.4 (7.1) | 34.4 (69.0)
  Cycle 1, Day 14 | 33.5 (47.4) | 0.0 (0.0) | 0.0 (0.0)

11. Secondary Outcome: Cmin of 5-FU
Time Frame: as for outcome 3
Population: PK analysis set population; number of participants analyzed (N): participants with evaluable data
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2
Number analyzed (Participants) | 2 | 9 | 10
ng/mL
  Cycle 1, Day 1 | 0.0 (0.0) | 0.0 (0.0) | 0.8 (2.5)
  Cycle 1, Day 14 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)

12. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) for SU, SU012662, and Total Drug (SU + SU012662)
Time Frame: Day 14 of Cycle 1 (predose and 2, 4, 6, 8, 10, and 24 hours postdose)
Population: PK analysis set population; number of participants analyzed (N): participants with evaluable data
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2
Number analyzed (Participants) | 2 | 9 | 10
hour (hr)
  Tmax SU011248 | 4.0 [4.0 to 4.0] | 8.0 [2.0 to 10.0] | 8.0 [4.0 to 10.0]
  Tmax SU012662 | 9.0 [8.0 to 10.0] | 8.0 [4.0 to 24.0] | 6.0 [0.0 to 10.0]
  Tmax total drug (SU011248+SU012662) | 4.0 [4.0 to 4.0] | 8.0 [2.0 to 10.0] | 6.0 [4.0 to 10.0]

13. Secondary Outcome: Tmax for CAP
Time Frame: as for outcome 3
Population: PK analysis set population; number of participants analyzed (N): participants with evaluable data
Measure: Median (Full Range); unit: hr
Arm/Group | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2
Number analyzed (Participants) | 2 | 9 | 10
hr
  Cycle 1, Day 1 | 4.3 [0.5 to 8.0] | 2.0 [0.5 to 3.0] | 0.5 [0.3 to 4.0]
  Cycle 1, Day 14 | 0.3 [0.3 to 0.3] | 2.0 [0.5 to 4.0] | 0.4 [0.0 to 3.0]

14. Secondary Outcome: Tmax for 5'DFCR
Time Frame: as for outcome 3
Population: PK analysis set population; number of participants analyzed (N): participants with evaluable data
Measure: Median (Full Range); unit: hr
Arm/Group | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2
Number analyzed (Participants) | 2 | 9 | 10
hr
  Cycle 1, Day 1 | 4.3 [0.5 to 8.0] | 2.0 [0.5 to 4.0] | 0.6 [0.5 to 4.0]
  Cycle 1, Day 14 | 0.4 [0.3 to 0.5] | 3.0 [0.9 to 4.0] | 0.5 [0.0 to 3.0]

15. Secondary Outcome: Tmax for 5'DFUR
Time Frame: as for outcome 3
Population: PK analysis set population; number of participants analyzed (N): participants with evaluable data
Measure: Median (Full Range); unit: hr
Arm/Group | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2
Number analyzed (Participants) | 2 | 9 | 10
hr
  Cycle 1, Day 1 | 4.5 [1.0 to 8.0] | 2.0 [0.5 to 4.0] | 0.8 [0.5 to 4.0]
  Cycle 1, Day 14 | 0.4 [0.3 to 0.5] | 3.0 [0.9 to 4.0] | 0.5 [0.0 to 3.0]

16. Secondary Outcome: Tmax for 5-FU
Time Frame: as for outcome 3
Population: PK analysis set population; number of participants analyzed (N): participants with evaluable data
Measure: Median (Full Range); unit: hr
Arm/Group | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2
Number analyzed (Participants) | 2 | 9 | 10
hr
  Cycle 1, Day 1 | 4.5 [1.0 to 8.0] | 2.0 [0.5 to 4.0] | 0.6 [0.3 to 4.0]
  Cycle 1, Day 14 | 0.4 [0.3 to 0.5] | 3.0 [0.5 to 4.0] | 0.5 [0.0 to 3.0]

17. Secondary Outcome: Terminal Elimination Half-Life (t1/2) for SU, SU012662, and Total Drug (SU + SU012662)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Day 14 of Cycle 1 (predose and 2, 4, 6, 8, 10, and 24 hours postdose)
Population: Not analyzed; t1/2 could not be accurately estimated due to the long t1/2 of SU and its active metabolite and due to short PK collection period of only 24 hrs.
Arm/Group | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2
Number analyzed (Participants) | 0 | 0 | 0

18. Secondary Outcome: t1/2 for CAP
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 3
Population: PK analysis set population; Number of participants analyzed (N): participants with evaluable data
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2
Number analyzed (Participants) | 1 | 1 | 9
hr
  Cycle 1, Day 1 | 0.3 (NA) — only 1 participant evaluated | 0.3 (NA) — only 1 participant evaluated | 0.4 (0.11)
  Cycle 1, Day 14 | 0.4 (NA) — only 1 participant evaluated | 0.5 (NA) — only 1 participant evaluated | 0.4 (0.12)

19. Secondary Outcome: t1/2 for 5'DFCR
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 3
Population: PK analysis set population; Number of participants analyzed (N): participants with evaluable data
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2
Number analyzed (Participants) | 1 | 6 | 10
hr
  Cycle 1, Day 1 | 0.7 (NA) — only 1 participant evaluated | 1.0 (0.4) | 0.8 (0.2)
  Cycle 1, Day 14 | 0.7 (NA) — only 1 participant evaluated | 1.1 (0.7) | 0.8 (0.1)

20. Secondary Outcome: t1/2 for 5'DFUR
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 3
Population: PK analysis set population; Number of participants analyzed (N): participants with evaluable data
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2
Number analyzed (Participants) | 1 | 5 | 10
hr
  Cycle 1, Day 1 | 0.7 (NA) — only 1 participant evaluated | 1.0 (0.4) | 0.7 (0.1)
  Cycle 1, Day 14 | 0.6 (NA) — only 1 participant evaluated | 1.0 (0.5) | 0.7 (0.1)

21. Secondary Outcome: t1/2 for 5-FU
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 3
Population: PK analysis set population; Number of participants analyzed (N): participants with evaluable data
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2
Number analyzed (Participants) | 1 | 2 | 9
hr
  Cycle 1, Day 1 | 0.8 (NA) — only 1 participant evaluated | 1.2 (0.8) | 0.6 (0.1)
  Cycle 1, Day 14 | 0.6 (NA) — only 1 participant evaluated | 1.1 (0.4) | 0.6 (0.1)

22. Secondary Outcome: Area Under the Curve From Time 0 to 24 Hours Postdose (AUC [0-24]) for SU, SU012662, and Total Drug (SU + SU012662)
Description: Area under the plasma concentration-time curve from time 0 to 24 hours postdose (0-24), also considered the AUC between doses at steady state.
Time Frame: Day 14 of Cycle 1 (predose and 2, 4, 6, 8, 10, and 24 hours postdose)
Population: PK analysis set population; Number of participants analyzed (N): participants with evaluable data
Measure: Mean (Standard Deviation); unit: nanogram hours per milliliter (ng*hr/mL)
Arm/Group | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2
Number analyzed (Participants) | 2 | 9 | 10
nanogram hours per milliliter (ng*hr/mL)
  AUC (0-24) SU011248 | 844 (155) [875 to 829] | 1420 (379) | 902 (230)
  AUC (0-24) SU012662 | 321 (254) | 524 (219) | 327 (64)
  AUC (0-24) total drug (SU011248+SU012662) | 1163 (407) [875 to 829] | 1944 (533) | 1230 (273)

23. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)]: CAP, 5'DFCR, 5'DFUR, and 5-FU
Description: AUC (0 - ∞) = Area under the plasma concentration versus time curve (AUC) from time zero (predose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Time Frame: Day 1 of Cycle 1 (0.25, 0.5, 1, 2, 3, 4, 8, and 10 hours postdose)
Population: PK analysis set population; Number of participants analyzed (N): participants with evaluable data; n: participants with evaluable data for specified category
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2
Number analyzed (Participants) | 1 | 7 | 10
ng*hr/mL
  CAP (n = 1, 4, 10) | 7480 (NA) — Only 1 participant evaluated | 2828 (215) | 8069 (3877)
  5'DFCR (n = 1, 7, 10) | 9200 (NA) — Only 1 participant evaluated | 8853 (1648) | 11467 (2476)
  5'DFUR (n = 1, 6, 10) | 7770 (NA) — Only 1 participant evaluated | 5703 (1295) | 9099 (2288)
  5-FU (n = 1, 5, 9) | 386 (NA) — Only 1 participant evaluated | 285 (119) | 489 (190)

24. Secondary Outcome: Area Under the Curve From Time Zero to 12 Hours [AUC (12)] for CAP, 5'DFCR, 5'DFUR, and 5-FU
Description: AUC (12) = Area under the plasma concentration versus time curve from time zero (predose) to the extrapolated time 12 hours postdose. It is obtained from AUC (0 - last) plus AUC (last - 12)
Time Frame: Day 14 of Cycle 1 (predose and 0.25, 0.5, 1, 2, 3, 4, 8, and 10 hours postdose)
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2
Number analyzed (Participants) | 1 | 7 | 10
ng*hr/mL
  CAP (n = 1, 4, 9) | 25435 (NA) — only 1 participant evaluated | 2663 (452) | 8865 (6533)
  5'DFCR (n = 1, 7, 10) | 15522 (NA) — only 1 participant evaluated | 7087 (1222) | 10091 (2847)
  5'DFUR (n = 1, 6, 10) | 15522 (NA) — only 1 participant evaluated | 4822 (1222) | 10291 (3675)
  5-FU (n = 1, 5, 10) | 1299 (NA) — only 1 participant evaluated | 353 (141) | 842 (403)

25. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for CAP
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Time Frame: Day 1 of Cycle 1 (0.25, 0.5, 1, 2, 3, 4, 8, and 10 hours postdose) and Day 14 of Cycle 1 (predose and 0.25, 0.5, 1, 2, 3, 4, 8, and 10 hours)
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2
Number analyzed (Participants) | 2 | 9 | 10
ng*hr/mL
  Cycle 1, Day 1 | 7555 (135) | 2899 (1580) | 7373 (4199)
  Cycle 1, Day 14 | 13532 (16648) | 3157 (1171) | 8213 (6432)

26. Secondary Outcome: AUClast for 5'DFCR
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Time Frame: as for outcome 25
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2
Number analyzed (Participants) | 2 | 9 | 10
ng*hr/mL
  Cycle 1, Day 1 | 12815 (5494) | 8028 (1963) | 11229 (2516)
  Cycle 1, Day 14 | 8614 (8477) | 6464 (1377) | 9776 (2868)

27. Secondary Outcome: AUClast for 5'DFUR
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Time Frame: as for outcome 25
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2
Number analyzed (Participants) | 2 | 9 | 10
ng*hr/mL
  Cycle 1, Day 1 | 8855 (1761) | 5658 (1237) | 8951 (2248)
  Cycle 1, Day 14 | 8500 (9192) | 4829 (1015) | 10017 (3637)

28. Secondary Outcome: AUClast for 5-FU
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Time Frame: as for outcome 25
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2
Number analyzed (Participants) | 2 | 9 | 10
ng*hr/mL
  Cycle 1, Day 1 | 355 (27) | 291 (95) | 506 (200)
  Cycle 1, Day 14 | 688 (802) | 350 (129) | 854 (390)

29. Secondary Outcome: Percentage of Participants With Objective Response
Description: Percentage of participants with an objective response-based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). CR defined as the disappearance of all target lesions. PR defined as ≥30 percent (%) decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: Baseline, Day 21 of every even-numbered cycle up to 15 months
Population: Efficacy analysis set population: all participants enrolled in the study who received at least 1 dose of study medication (SU011248).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SU 37.5 mg, CIS 60 mg/m^2, CAP 1600 mg/m^2 | SU 37.5 mg, CIS 60 mg/m^2, CAP 2000 mg/m^2 | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2
Number analyzed (Participants) | 6 | 7 | 15 | 23 | 3 | 22
percentage of participants | 16.7 [0.4 to 64.1] | 42.9 [9.9 to 81.6] | 46.7 [21.3 to 73.4] | 43.5 [23.2 to 65.5] | 0 [0.0 to 70.8] | 45.5 [24.4 to 67.8]

30. Secondary Outcome: Duration of Response (DR)
Description: DR defined as time from start of first documented objective tumor response (CR or PR) to first documented objective tumor progression or death due to any cause, whichever occurs first.
Time Frame: Baseline up to Month 15
Population: Efficacy analysis set population; No participants in the SU 37.5 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2 reporting group analyzed; all had stable disease during specified time frame
Measure: Median (Full Range); unit: months
Arm/Group | SU 37.5 mg, CIS 60 mg/m^2, CAP 1600 mg/m^2 | SU 37.5 mg, CIS 60 mg/m^2, CAP 2000 mg/m^2 | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2
Number analyzed (Participants) | 1 | 3 | 7 | 10 | 10
months | 14.1 [14.1 to 14.1] | 6.3 [6.0 to 10.9] | 10.5 [4.4 to 28.1] | 5.9 [2.8 to 12.8] | 6.3 [2.5 to 25.5]

31. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS defined as time from the first dose of study treatment to the first documentation of objective tumor progression or to death due to any cause, whichever occurs first.
Time Frame: Baseline up to Month 15
Population: Efficacy analysis subset of population of participants who had an event
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | SU 37.5 mg, CIS 60 mg/m^2, CAP 1600 mg/m^2 | SU 37.5 mg, CIS 60 mg/m^2, CAP 2000 mg/m^2 | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2
Number analyzed (Participants) | 6 | 6 | 11 | 16 | 3 | 17
months | 3.2 [2.7 to 9.3] | 6.6 [2.5 to 8.0] | 6.4 [4.3 to 13.9] | 8.0 [4.7 to 9.4] | 2.8 [2.3 to 11.7] | 5.5 [4.7 to 10.1]

ADVERSE EVENTS:
Description: The same event may appear as an adverse event (AE) and serious AE (SAE). However, what is presented are distinct events. An event may be serious in 1 participant and nonserious in another, or 1 participant may have experienced both a serious and nonserious event during the study. Event assessments were made on a regular schedule as per protocol.
Arm/Group | SU 37.5 mg, CIS 60 mg/m^2, CAP 1600 mg/m^2 | SU 37.5 mg, CIS 60 mg/m^2, CAP 2000 mg/m^2 | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 | SU 37.5 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2 | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2
Serious Adverse Events (participants affected / at risk) | 1/6 | 2/7 | 8/15 | 8/23 | 0/3 | 5/22
Other Adverse Events (participants affected / at risk) | 6/6 | 7/7 | 15/15 | 23/23 | 3/3 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SU 37.5 mg, CIS 60 mg/m^2, CAP 1600 mg/m^2 (N=6) | SU 37.5 mg, CIS 60 mg/m^2, CAP 2000 mg/m^2 (N=7) | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 (N=15) | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 (N=23) | SU 37.5 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2 (N=3) | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2 (N=22)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Duodenal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 2 | 0 | 1
Sudden death (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Infectious peritonitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SU 37.5 mg, CIS 60 mg/m^2, CAP 1600 mg/m^2 (N=6) | SU 37.5 mg, CIS 60 mg/m^2, CAP 2000 mg/m^2 (N=7) | SU 25 mg, CIS 80 mg/m^2, CAP 2000 mg/m^2 (N=15) | SU 37.5 mg, OXA 110 mg/m^2, CAP 1600 mg/m^2 (N=23) | SU 37.5 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2 (N=3) | SU 25 mg, OXA 110 mg/m^2, CAP 2000 mg/m^2 (N=22)
Anaemia (Blood and lymphatic system disorders) | 4 | 4 | 9 | 8 | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 3 | 3 | 0 | 1 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 5 | 6 | 15 | 18 | 2 | 18
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 6 | 10 | 16 | 2 | 8
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 1 | 4 | 1 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 1 | 5 | 1 | 4
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 4 | 7 | 6 | 1 | 10
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2 | 3 | 9 | 0 | 6
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 4 | 3 | 7 | 8 | 0 | 5
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 6 | 12 | 0 | 11
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 6 | 5 | 1 | 3
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 6 | 12 | 17 | 2 | 17
Rectal tenesmus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 5 | 3 | 8 | 10 | 1 | 7
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 4 | 5 | 8 | 0 | 7
Asthenia (General disorders) | 0 | 1 | 1 | 3 | 0 | 1
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 1 | 2
Chest pain (General disorders) | 1 | 0 | 1 | 1 | 0 | 1
Chills (General disorders) | 0 | 0 | 2 | 2 | 0 | 0
Face oedema (General disorders) | 1 | 2 | 0 | 7 | 1 | 2
Fatigue (General disorders) | 6 | 6 | 5 | 9 | 1 | 8
Mucosal inflammation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oedema (General disorders) | 1 | 0 | 1 | 0 | 0 | 2
Oedema peripheral (General disorders) | 1 | 1 | 0 | 0 | 0 | 2
Pain (General disorders) | 1 | 0 | 0 | 2 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 4 | 0 | 2
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 2 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 0 | 2 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 5 | 2 | 2
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 3 | 1 | 0 | 2
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 2 | 2 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 4 | 1 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 5 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 2 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 1
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Platelet count (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 3 | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 6 | 11 | 15 | 3 | 13
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 2 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 3 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 3 | 0 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 2 | 0 | 6
Dysgeusia (Nervous system disorders) | 1 | 1 | 1 | 7 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 3 | 4 | 0 | 5
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 2 | 6 | 1 | 8
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1 | 3 | 6 | 0 | 5
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 1 | 4 | 2 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 1 | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 3 | 0 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 2 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 4 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1 | 2 | 1 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 4 | 8 | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 2 | 0 | 3
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 1 | 2 | 1 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pericoronitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.